CLINICAL TRIAL: NCT05651425
Title: A Retrospective, Multicenter, Controlled Clinical Trail: to Evaluate the Efficiency and Safety of Intracranial Aneurysm Assistive Software in the Preoperative Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: QX2022-011-02
Record Dates: First submitted 2022-11-23; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysm; intravascular coiling embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Clinical data of all patients enrolled in our trial are preserved in CRF format, and CTA data are preserved in DICOM format.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgeon-independent group: the coiling diameter is predicted by experienced surgeon alone.
- surgeon-software-assistant group: the coiling diameter is predicted by experienced surgeon with software assistant.

SUMMARY:
the goal of this clinical trail is to evaluate the efficiency and safety of intracranial aneurysm assistive software in the preoperative assessment. The trail is designed as retrospective, multicenter, controlled clinical trail. Collecting probable cases images retrospectively according to inclusion criteria and exclusion criteria strictly. Controlling bias strictly, to make sure the efficiency and safety of intracranial aneurysm assistive software is evaluated reliably and precisely. In our trail, software-assisstant planning controls against experienced-surgeon-independent planning，which aims to avoid bias effictively and eliminate non-test interferences.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-80y, no gender limitation.
2. non-ruptured intracranial saccular aneurysm with specific intracranial CTA images; Target aneurysm has performed intravascular coiling treatment.
3. intracranial aneurysm diameter range from 3mm to 10mm.
4. the shape of aneurysm is regular without daughter sac or more than 2 lobulations.

Inclusion criteria of images:

1. the number of detector rows of Computed Tomography(CT) is more than 16 rows.
2. slice thickness ≤ 0.625mm, whole-brain image is considered.
3. Both plain scan sequences and enhancer sequence are required.

Exclusion Criteria:

1. combined with cerebral hemorrhage;
2. combined with cerevascular malformation or cerebral occupying lesion;
3. fusiform aneurysm or dissection aneurysm;
4. significant proximal stenosis of parent artery;
5. intracaverous internal carotid artery aneurysm;
6. target aneurysm has been performed flow-diverter stents treatment.

Exclusion criteria of images:

1. none DICOM format;
2. quality score less than 3 scores;
3. metal artifacts existance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
concordance rate | accessment time point : immediately after computational coiling diameter assessment finished.
  the optimal coiling diameter used in surgery is considered as "gold standard". The concordance rate is defined as computational suitable coiling diameter in test group differs gold standard less than ±1mm.
  concordance rate=the number of concordance matched/totle enrolled number*100%

SECONDARY OUTCOMES:
coincidence rate | accessment time point: immediately after computational coiling diameter assessment finished.
  the optimal coiling diameter used in surgery is considered as "gold standard". The coincidence rate is defined as computational suitable coiling diameter in test group is less than gold standard.
  coincidence rate= the number meets coincidence requirement /totle enrolled *100%

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China